CLINICAL TRIAL: NCT00973739
Title: Phase II Study of Lapatinib in Children and Adults With Neurofibromatosis Type 2(NF2) and NF2-related Tumors
Brief Title: Lapatinib Study for Children and Adults With Neurofibromatosis Type 2 (NF2) and NF2-Related Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0328
Record Dates: First submitted 2009-09-03; First posted 2009-09-09 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Neurofibromatosis 2; Vestibular Schwannoma
Keywords: NF-2; NF-2 related tumors; Schwannoma, Acoustic, Bilateral; schwannomas; Neurilemmoma of other cranial and peripheral nerves; NF2 related benign intracranial tumors including; NF2 related meningiomas; NF2 related ependymomas; NF2 related spinal neurofibromas; NF2 related gliomas
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic; Neurilemmoma | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib (Experimental): Lapatinib PO dosed according to age:
  Children/adolescents (less than 18 years of age): 1,800 mg/m2/day PO divided into twice daily doses, to a maximum of 750 mg PO twice daily
  Adults (18 years of age or older): 1,500 mg PO once daily
  Lapatinib is available in 250 mg tablets only. For pediatric dosing, the total daily dose will be rounded up or down to the nearest 250 mg increment.
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — Lapatinib is dosed according to age. Lapatinib is available in 250 mg tablets only. For pediatric dosing, the total daily dose will be rounded up or down to the nearest 250 mg increment.
  Children/adolescents (<18 years of age): 1,800 mg/m2/day PO divided into twice daily doses, to a maximum of 750 mg PO (3 tablets twice daily)
  Adults (>=18 years of age): 1,500 mg PO (6 tablets once daily)
  Duration: Up to 12 months, depending on treatment response.
  Other Names: Tykerb

SUMMARY:
The purpose of this study is to determine if Lapatinib has any effect on tumors found in patients with Neurofibromatosis Type 2 (NF2). NF2 is a condition that mainly affects the skin and nervous system. It causes non-cancerous tumors (which are known as neuromas) to grow on the nerves around a person's body. Some signs of NF2 include a gradual loss of hearing and tumors growing on the skin, the brain and the spinal cord which can lead to complications.

Lapatinib is an oral drug that is approved by Food and Drug Administration (FDA) for other types of tumors, it is not approved by the FDA for treatment of NF2 related tumors. The investigators know a lot about how well it is tolerated, but the investigators do not know if it is effective in treating your condition, therefore it is considered to be an investigational medication. This study will test whether Lapatinib may shrink tumors commonly found in patients with NF2 or stop them from growing. This will help us to decide if Lapatinib should be used to treat NF2 patients in future. Lapatinib is a drug that has been used for over 10 years to treat various forms of cancer. It has not been studied for the treatment of tumors in NF2 patients.

DETAILED DESCRIPTION:
In this trial, we propose to assess the objective response rates to Lapatinib in patients with NF2-related tumors. Lapatinib is a commercially available inhibitor of ErbB2 and EGF. Data suggests that abnormal signaling via EGFR and ErbB2 is a major contributor to tumor growth and progression in both sporadic and NF2-related VS and that inhibition of this signaling pathway can result in decreased tumor growth.

Demonstrating that Lapatinib produces an objective response to reduce tumor volume or stabilize disease will provide additional treatment options for NF patients with multiple tumor growth. For patients with VS we expect to see ≥ 10 dB improvement in PTA and/or improvement in SDS, compared to the audiogram at initiation of treatment. Currently there are no available treatment options for NF2 patients with multiple tumors. Depending on tumor cell type, lapatinib has cytostatic or cytotoxic antitumor effects, and in a recent study assessing the biological effects of Lapatinib on the associated molecular pathways and tumor growth in patients with solid tumors, a correlation was seen between tumor response and pre-treatment levels of (phosphor)-ErbB2 and (phosphor)-ERK1/2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 4 years of age.
2. Patients must meet diagnostic criteria for NF2 and at least one volumetrically measured NF2-related brain or spinal tumor with radiographic evidence of progression over the past 12 months, designated as the primary target OR volumetrically measurable VS with ipsilateral progressive hearing loss over the past 12 months, designated as the primary target tumor.
3. Significant hearing loss criteria for enrollment.
4. Karnofsky (PS) OR Lansky 50-100% (>16 years of age)
5. Absolute neutrophil count ≥ 1,000/mm3 g/dL
6. Hemoglobin ≥ 8 g/dL
7. Creatinine ≤ 1.5 times upper limit of normal (ULN) OR corrected glomerular filtration rate ≥ 70 ml/min
8. Bilirubin ≤ 1.5 times ULN
9. ALT ≤ 2.5 times ULN
10. Fully recovered from acute toxic effects of any prior chemotherapy, biological modifiers or radiotherapy.
11. Steroids are allowed for progressive symptoms but patient must be on a stable dose for at least 1 week prior to study entry.
12. Any neurologic deficits must be stable for ≥ 1 week.
13. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test. The anti-proliferative activity of this experimental drug may be harmful to the developing fetus.
14. Normal cardiac left ventricular ejection fraction (LVEF) by transthoracic echocardiogram.
15. Able to provide written informed consent (or consent by parent/legal guardian for minors)

Exclusion Criteria:

1. Patients with serious concurrent infection or medical illness.
2. Neurological deficits that are rapidly progressing.
3. Patients who are pregnant or breast-feeding.
4. Anti-tumor therapy within 4 weeks prior to enrollment.
5. Radiation therapy within 2 months prior to enrollment.
6. Prior therapy with agents targeting EGFR or ErbB2.
7. Any surgery within 4 weeks prior to enrollment.
8. Significant gastrointestinal disorder(s)
9. Known cardiac disease
10. Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Patients who have been free of disease (any prior malignancy) for more than five years are eligible for this study.
11. Patients cannot have received cytochrome P450-inducing anticonvulsants (EIADs; e.g., phenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine) or similar agents (e.g., rifampin) or P450-inhibiting agents (Ketoconazole, Itraconazole, Clarithromycin, Atazanavir, Indinavir, Nefazodone, Nelfinavir, Ritonavir, Saquinavir, Telithromycin, Voriconazole)

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias A Karajannis, MD, MS, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-one patients were enrolled between October 2009 and March 2011 at New York University Medical Center.
Groups:
- Lapatinib: Lapatinib will be administered
Period: Overall Study
Arm/Group | Lapatinib
Started | 21
Completed | 17
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Estimated Volumetric Progression Free Survival at 12 Months
Description: Measurements were taken every three months, up to one year. Estimated volumetric progression free survival (PFS) was measured from date of enrollment to date of volumetric progression. PFS was analyzed using the Kaplan-Meier method in terms of overall PFS (volumetric or hearing progression), volumetric progression, and hearing progression.
  Point estimates for PFS with 95% confidence intervals (CIs) were calculated from Kaplan-Meier curves.
Time Frame: Every three months for one year
Population: This analysis is based on the 17 evaluable patients.
Measure: Mean (95% Confidence Interval); unit: Liklihood of PFS at 12 months
Arm/Group | Lapatinib
Number analyzed (Participants) | 17
Liklihood of PFS at 12 months | 70.6 [43.1 to 86.6]

2. Secondary Outcome: Estimated Volumetric Progression Free Survival for Hearing at 12 Months
Description: Measurements were taken every three months, up to one year. Estimated volumetric progression free survival (PFS) was measured from date of enrollment to date of hearing progression. PFS was analyzed using the Kaplan-Meier method in terms of overall PFS (volumetric or hearing progression), volumetric progression, and hearing progression.
  Point estimates for PFS with 95% confidence intervals (CIs) were calculated from Kaplan-Meier curves.
Time Frame: Every three months for one year
Population: This analysis is based on the 17 evaluable patients.
Measure: Mean (95% Confidence Interval); unit: Liklihood of PFS at 12 months
Arm/Group | Lapatinib
Number analyzed (Participants) | 17
Liklihood of PFS at 12 months | 88.9 [43.3 to 98.4]

3. Secondary Outcome: Participants Experiencing Grades 1 or 2 Toxicities (CTCAE)
Description: Toxicity was assessed throughout the study, up to one year.
Time Frame: Baseline through one year
Measure: Number; unit: participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 21
participants | 21

4. Secondary Outcome: Participants Experiencing Grade 3 Toxicities (CTCAE)
Description: Toxicity was assessed throughout the study, up to one year.
Time Frame: Baseline through one year
Measure: Number; unit: participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 21
participants | 1

ADVERSE EVENTS:
Arm/Group | Lapatinib
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib (N=21)
Vasovagal syncope (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Decreased bicarbonate (Metabolism and nutrition disorders) | 5 (5)
Dermatology/Skin (Other) (Skin and subcutaneous tissue disorders) | 19 (19)
Diarrhea (Gastrointestinal disorders) | 15 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1)
Hemorrhage - rectum (stools) (Gastrointestinal disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
Increased ALT (Investigations) | 4 (4)
Increased AST (Investigations) | 7 (7)
Increased PTT (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Keratitis (Eye disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Memory Impairment (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Numbness L-S area (Nervous system disorders) | 1 (1)
Pain-Other (General disorders) | 8 (8)
Pericardial effusion on echocardiogram (Cardiac disorders) | 1 (1)
Possible ectopic atrial bradycardia on EKG (Cardiac disorders) | 1 (1)
Premature supraventricular complexes on EKG (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 2 (2)
Stomatitis (oral cavity ulceration) (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No